CLINICAL TRIAL: NCT06374667
Title: The Efficacy and Safety of Y-3 Intracalvariosseous Injection Bypassing Blood-brain Barrier Versus Intravenous Injection in the Treatment of Acute Large Hemispheric Infarction（SOLUTION-2）
Brief Title: The Efficacy and Safety of Y-3 Intracalvariosseous Injection Versus Intravenous Injection in the Treatment of Acute Large Hemispheric Infarction
Acronym: SOLUTION-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: yilong Wang (Other)
Responsible Party: Sponsor-Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024-071-02
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Acute Ischemic; Blood-Brain Barrier
Keywords: large hemispheric infarction; Y-3; postsynaptic density protein 95 inhibitor; BBB-bypassing route; brain drug delivery; intracalvariosseous injection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICO injection group (Experimental): Y-3 ICO injection (dose was given as 32 ug/kg) once a day for 3 consecutive days, as well as standard treatment and management according to the related guidelines.
  Interventions: Procedure: Y-3 ICO injection; Other: Conventional treatment
- intravenous injection group (Active Comparator): Y-3 intravenous injection(dose was given as 40mg + 250ml normal saline), as well as standard treatment and management according to related guidelines.
  Interventions: Drug: Y-3 intravenous injection; Other: Conventional treatment

INTERVENTIONS:
Procedure: Y-3 ICO injection — Patients included will be given skull outer plate drilling surgery and Y-3 ICO injection under local anesthesia and sedation. The injection will be given for 3 consecutive days.
  Arms: ICO injection group
Drug: Y-3 intravenous injection — Patients included will be given Y-3 intravenous injection for 7 consecutive days.
  Arms: intravenous injection group
Other: Conventional treatment — standard treatment and management according to related guidelines during the entire treatment period

SUMMARY:
A pilot study confirmed the feasibility and safety of neuroprotectant Y-3 intracalvariosseous(ICO) injection in patients with malignant middle cerebral artery infarction (mMCAI), showing a trend in improving 90-day functional scores compared to conventional treatment. The aim of this trial is to further investigate the efficacy and safety of ICO injection of Y-3 compared to intravenous injection in patients with acute large hemispheric infarction(LHI) who has contraindications of reperfusion therapy or have got poor reperfusion therapy outcomes.

DETAILED DESCRIPTION:
The mortality rate of large hemispheric infarction(LHI) is up to 40%-60%, while current available treatment is limited. Mainstream therapeutics include endovascular reperfusion therapy and decompressive craniectomy. But endovascular-reperfusion has limits such as short time window and hemorrhagic transformation risk, while decompressive craniectomy can reduce mortality but not infarct volume. Curative effect of intravenous injection of neuroprotective drugs is severely limited because of the blood-brain barrier. Microchannels connecting the skull bone marrow and dura may be effective drug delivery shortcuts bypassing the blood-brain barrier. Cytoprotective drug Y-3 affects dual aspects of ischemic cascade by disrupting both function of the synaptic folding post-synaptic density protein 95 (PSD-95), as well as α2-γ⁃Aminobutyric acid type A receptor (α2-GABAAR) agonist. Phase I and Phase II clinical trials have confirmed the safety and efficacy of intravenous infusion of Y-3 in treating cerebral infarction, with the optimal dosage being 40mg. Preclinical testing proved that ICO injection of Y-3 solution 24h post rat permanent middle cerebral artery infarction reduced rat infarction volume and improved neurological function.

SOLUTION-2 is a multicentered, prospective, randomized, open-label, blinded end-point (PROBE) study

The purpose of this study is to investigate the efficacy and safety of ICO injection of Y-3 compared to intravenous injection in acute LHI patients with contraindications of reperfusion therapy or poor outcomes.

Patients will be randomly assigned to one of the following 2 groups at 1:1 ratio.

ICO injection group: Y-3 ICO injection (dose was given as 32 ug/kg) once a day for 3 consecutive days, as well as standard treatment and management according to the related guidelines.

intravenous injection group: Y-3 intravenous injection(dose was given as 40mg + 250ml normal saline), as well as standard treatment and management according to related guidelines.

Face to face interviews will be made on baseline, 4±1 days after randomization, 8±1 days after randomization, 14±1 days after randomization or discharge day, and 90 days , 1year± 14 days after randomization.

The primary efficacy outcomes is the modified Rankin Scale（mRS） 0-3 points at 90±7 days. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by Institutional Review Board (IRB) and Ethics Committee (EC) in Being Tiantan hospital, Capital Medical University.

ELIGIBILITY:
Inclusion Criteria:

* 18≤Age≤80 years;
* First stroke or complete self-care before the onset of current stroke (mRS 0-1);
* Administration of drugs can be completed within 24h of the onset of signs and symptoms of neurological deficits (in patients with wake-up strokes or unwitnessed strokes, the time of onset is defined as the time of last normal presentation);
* Clinical symptoms, signs and imaging diagnosis of cerebral infarction in the area supplied by the middle cerebral artery, together with the following features:

  1. 16≤ NIHSS ≤32 points, and the sum of the scores of motor arm and motor leg is ≥6;
  2. Imaging suggestive of core infarct area: apparent diffusion coefficient (ADC) values <620×10^-6mm^2/s lesion volume on magnetic resonance imaging (MRI) diffusion-weighted imaging (DWI) sequences or cerebral blood flow (CBF) <30% of volume 70-300 ml on computed tomography perfusion imaging (CTP) or an Alberta Stroke Program Early CT Score (ASPECTS) of 0-6, with inconsistent findings, the investigator is required to make a reasoned judgement by taking into account all the information (scanning time, the imaging method that best responds to the size of infarct, etc.) and record it.
* NIHSS score not improving or progressing after reperfusion therapy and total score still ≤32.
* Informed consent signed

Exclusion Criteria:

* Complications with other cerebrovascular diseases meet one of the following conditions:

  1. Complicated with acute cerebral hemorrhage and subarachnoid hemorrhage;
  2. Complicated with acute posterior circulation cerebral infarction or severe posterior circulation stenosis (>70%);
  3. Or imaging suggests that the area of cerebral infarction is involved bilaterally;
  4. The cause of the TOAST classification was considered as intracranial artery dissection, vasculitis, moyamoya disease and other etiological types.
* Hemorrhage transformation in the infarction area, hematoma area ≥30% of the infarction area, and has obvious space-occupying effect;
* Presence of clinical signs of brain herniation formation, e.g., unilateral or bilateral pupil dilation and fixation; cerebral oedema-associated loss of consciousness (NIHSS 1a > 2 points), or other loss of brainstem reflexes in the judgement of the investigator, caused by cerebral oedema or cerebral herniation formation; or other signs of instability of vital signs that are difficult to control;
* Craniotomy decompression was planned before randomization;
* Refractory hypertension (systolic > 200mmHg or diastolic > 110mmHg) or hypotension (systolic < 70mmHg or diastolic < 50mmHg) that is difficult to control with medication;
* Abnormal blood glucose before randomization (random venous blood glucose < 2.8mmol/L or > 23mmol/L);
* Presence of significant abnormal liver function markers or renal function markers prior to randomization;
* Note: Severe liver function abnormalities were defined as serum alanine aminotransferase (ALT), or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN). Significant renal insufficiency is defined as eGFR less than 60 mL/min/1.73 m² (eGFR, calculated using the CKD-EPI formula)
* Acute ST-elevation myocardial infarction (MI) and/or decompensated heart failure (meeting the New York College of Cardiology (NYHA) Heart function grades III and IV) within the past 3 months;
* Presence of contraindications to intracalvariosseous injection, e.g., skull fracture in the last 3 months, skull infection, subdural/extradural hematoma, subcutaneous hematoma, skin or subcutaneous infection of the scalp, poorly displayed skull bone marrow niches；
* Bleeding tendencies considered by the investigators to be detrimental to the procedure include, but are not limited to, platelet counts < 100×10^9/L, and the presence of clotting disorders such as hemophilia；
* Presence of severe or very severe anemia (hemoglobin <60 g/L) at randomization；
* Patients with severe respiratory diseases (severe chronic obstructive pulmonary disease, respiratory failure, etc.) should be corrected by intubation, tracheotomy, or ventilator;
* The subjects were considered to have developed clinically significant serious infections, including severe local infections or systemic infections;
* Diagnosed severe degenerative diseases of the central nervous system such as Alzheimer's Disease (AD), Parkinson's Disease (PD), and severe dementia of all causes, or psychiatric disorders (e.g., schizophrenia, depression, etc.);
* Subjects with a life expectancy of less than 3 months due to conditions not considered current by the investigators, such as tumors;
* Known allergy to any component of investigational process therapy drugs and contrast agents;
* Subjects who are pregnant, breastfeeding or have the possibility of becoming pregnant or plan to become pregnant;
* Subjects are unable to comply with trial protocols or follow-up requirements;
* Other circumstances deemed by the investigators to be unsuitable for enrollment (registration of reasons for inability to enroll is required);
* Have participated in other interventional clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
90-day favorable clinical outcome | 90±7 days after randomization
  Favorable clinical outcome defined as a dichotomized mRS 0-3 outcome The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead

SECONDARY OUTCOMES:
Change of infarct volume from baseline to 8-day | baseline，8±1 days after randomization
  The infarct volume is determined on a diffusion-weighted MRI map based on an ADC threshold of less than 620 ×10^-6mm^2/s or on CTP image with rCBF<30%
Neurofunctional deficit defined as the National Institutes of Health Stroke Scale (NIHSS) . | 8±1 days after randomization，14±1 days after randomization，90±7 days after randomization
  NIHSS is a standardized neurological examination score that is a valid and reliable measure of disability and recovery after acute stroke. Scores range from 0 to 42, with higher scores indicating increasing severity.
Patients with symptoms improvement from baseline to 14-day | baseline，14±1 days after randomization
  Symptoms improvement defined as the NIHSS scores improved by 4 points from baseline to 14-day
Rate of decompressive hemicraniectomy | 90±7 days after randomization
  Rate of decompressive hemicraniectomy
Depression scale scores at 90-day | 90±7 days after randomization
  Depression scale scores including Stroke Aphasic Depression Questionnaire-Hospital Version(SADQ-H) and Aphasia Depression Rating Scale(ADRS)
Proportion of combined adverse events at 90-day | 90±7 days after randomization
  Combined adverse events defined as mRS 4-5, decompressive craniotomy, vascular death
90-day modified Rankin Scale | 90±7 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead

OTHER OUTCOMES:
1-year favorable clinical outcome | 1 year±14 days after randomization
  Favorable clinical outcome defined as a dichotomized mRS 0-3 outcome The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead
1-year modified Rankin Scale | 1 year±14 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead
1-year anterior circulation Alberta Stroke Program Early CT Score | 1 year±14 days after randomization
  Alberta Stroke Program Early CT Score（ASPECTS）, a scale from 0-10 to measure infarct size, with lower scores reflecting larger infarcts

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, PhD，MD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (6):
- China (6):
  - The first affiliated hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Heibei
  - Tangshan Municipal Worker's Hospital, Tangshan, Heibei
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Tianjin Huanhu hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang N, Zhang M, Yang M, Liu W, Liu W, Ou Y, Zhou M, Wang X, Sun Z, Pan Y, Wang Y, Wang Y. Efficacy and safety of Y-3 intracalvariosseous injection versus intravenous injection in the treatment of acute large hemispheric infarction (SOLUTION-2): rationale and design of a multicentre, prospective, randomised, open-label, blind endpoint (PROBE) trial. Stroke Vasc Neurol. 2025 Jun 3:svn-2024-004011. doi: 10.1136/svn-2024-004011. Online ahead of print. PMID 40461153